CLINICAL TRIAL: NCT06405984
Title: Trans-Abdominal Fetal Pulse Oximetry - An Early Feasibility Study
Brief Title: Trans-Abdominal Fetal Pulse Oximetry - EFS-IDE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Raydiant Oximetry, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP2340; R44HD094486 (NIH)
Record Dates: First submitted 2024-04-03; First posted 2024-05-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Fetal Hypoxia; Fetal Distress; Fetal Conditions; Fetal Complications; Labor Fetal Anoxia; Labor (Obstetrics)--Complications; Oxygen Deficiency
Keywords: fetal hypoxia; fetal distress; oxygen deficiency; labor fetal anoxia
MeSH Terms: conditions — Fetal Hypoxia; Fetal Distress; Hypoxia

STUDY DESIGN:
Intervention Model Description: This is a single-arm, device feasibility study, based on convenience sampling.
Masking Description: Although it is known what devices are used, all personnel on the investigative team will be masked to fetal oxygenation levels during data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Laboring Women (Experimental): Women in labor who have consented to participation in the study.
  Interventions: Device: Fetal Oxygenation Measurements

INTERVENTIONS:
Device: Fetal Oxygenation Measurements — The Lumerah device, and Oxiplex ISS will be positioned on the maternal abdomen in various locations depending on the sonographic evaluation. The transvaginal sensor will be placed after rupture of the maternal membranes and appropriate descent of the fetus.This study is for data collection purposes only. Neonates of this study arm will also be monitored with the Oxiplex ISS system. This study is for data collection purposes only.

SUMMARY:
The Lumerah System, developed and manufactured by Raydiant Oximetry, Inc., is a non-invasive fetal pulse oximeter that measures fetal arterial oxygen saturation using safe, non-invasive, transabdominal near-infrared spectroscopy. The Lumerah System is intended as an adjunct to cardiotocography. In this study, women in labor will also be simultaneously monitored with a re-engineered version of the previously approved transvaginal oximeter sensor connected to a Nellcor N-400 fetal oximetry monitor for the purposes of device development. The data obtained from the transabdominal sensor and the transvaginal sensor will be used for research purposes only and will not be used to guide or alter patient management.

DETAILED DESCRIPTION:
This is a prospective, interventional, open-label, Early Feasibility Study Investigational Device Exemption (EFS-IDE). The Principal Investigator or research team member will consult a list of eligible patients based on predicted delivery dates and scheduled inductions. Women who are planning to undergo labor will be approached regarding this study. The study involves measurement of the fetal pulse signal with the investigational device, Lumerah, during labor. Lumerah is an investigational fetal pulse oximeter that measures fetal arterial oxygen saturation using safe, non-invasive, transabdominal near-infrared spectroscopy. The Lumerah device is intended as an adjunct to cardiotocography by detecting fetal oxygen deprivation that is both life-threatening to the fetus and can lead to the irreversibly debilitating consequences of newborn metabolic acidosis. The subjects will first undergo sonographic evaluation to assess distance from maternal skin to fetal tissue and to confirm fetal presentation and position during labor. The results of the sonographic measurements might influence the enrollment suitability of the subject as well as the placement of the Investigational device. The Oxiplex TS device, a non-ionizing laser system that provides researchers with valuable information regarding maternal optical tissue properties, will also be used. Once the membranes are ruptured, the investigator's team will use a Nellcor N-400 System with a sterile, single-use transvaginal sensor for data collection only. The outcomes of the fetal oxygenation measurements are masked; only the Sponsor is aware of the measurements. Therefore, no clinical decisions will be made based on the information derived from any of the devices used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable to provide informed consent
2. Age > 18 years
3. < 4 cm between maternal skin and fetal skin (determined by ultrasound)
4. Gestational age > 36 weeks
5. Singleton pregnancy
6. Vertex presentation
7. Active labor
8. Category I and Category II tracings, and
9. Ruptured amniotic sac with cervical dilation of >2 cm and a station of -2 or lower

Exclusion Criteria:

1. Age < 18 years
2. Gestational age < 36 weeks
3. Multiple gestation
4. Nonvertex fetal presentation
5. Suspected vasa previa
6. Latent labor
7. Category III CTG tracing (i.e., need for immediate delivery)
8. Fetal anomalies and/or chromosomal disorders
9. Chorioamnionitis
10. Placenta Previa
11. History of HIV, Genital Herpes, or other infection precluding transvaginal monitoring
12. Unable to provide informed consent (e.g., cognitively impaired)
13. > 4 cm fetal depth (determined by Ultrasound),
14. Low anterior placenta, or
15. Any condition (temporary or permanent) in which the investigator deems the patient unsuitable for the study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study applies to women in labor
Enrollment: 35 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of monitoring fetal signals. | During labor for up to 6 hours
  Prototype device feasibility of detecting reflected optical signals at different wavelengths ("colors") from the fetus
Safety of the prototype device | Up to 72 hours post partum
  Rate of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Sentara Norfolk General - Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
This is a data collection study whereby data will be used for device development purposes. There is no plan to share these data with other researchers.